CLINICAL TRIAL: NCT04598386
Title: The Effect of AMP Human Sodium Bicarbonate Lotion on Hydration (AMPlify Human Hydration Study)
Brief Title: The Effect of AMP Human Sodium Bicarbonate Lotion on Hydration
Acronym: AMPlify
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: AMP Human; Park City, UT (Unknown); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Douglas J Casa, Principal Investigator, University of Connecticut
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H20-0100
Record Dates: First submitted 2020-10-07; First posted 2020-10-22 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Fluid Retention; Fluid Loss; Sodium Retention; Cognitive Change; Heat Exposure; Hyperhydration; Electrolyte and Fluid Balance Conditions
Keywords: Sodium Bicarbonate; Topical Lotion
MeSH Terms: conditions — Hypernatremia; Water Intoxication

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PR Lotion Topical Solution (Experimental): Approximately 50 grams of PR Lotion will be applied by the participants to their upper extremities (arms) in addition to their neck, upper back, chest, and midsection if necessary. This lotion will be applied once during the 4th of session of their PR Lotion Phase and will remain on the skin for approximately 4.5 hours.
  Interventions: Other: PR Lotion - AMP Human Performance
- Placebo Lotion Topical Solution (Placebo Comparator): Approximately 50 grams of the Placebo Lotion will be applied by the participants to their upper extremities (arms) in addition to their neck, upper back, chest, and midsection if necessary. The only difference in ingredients for this Placebo Lotion will be the exclusion of the sodium bicarbonate ingredient. This lotion will be applied once during the 4th of session of their Placebo Lotion Phase and will remain on the skin for approximately 4.5 hours.
  Interventions: Other: Placebo Lotion

INTERVENTIONS:
Other: PR Lotion - AMP Human Performance — Sodium Bicarbonate Topical Solution. For use of the PR Lotion solution, consumers are instructed to apply the lotion to areas of the body that have been identified as most likely to use during their activity (i.e. calves and thighs for runners, shoulders and forearms for swimmers, etc.). Moreover, the product can be applied up to 2 hours prior to beginning a workout or event with one use supporting a 4-6 hour workout. AMP Human has also verified the safety of their product as being well tolerated in consumers >2 years of age unless there is a known allergy to an ingredient on the label. Moreover, to the company's knowledge no side effects have been reported per the SAFETY Section at https://amphuman.com/pages/faq.
  Other Names: NDC Code: 72358-101-01; NDC Code: 72358-101-02; NDC Code: 72358-101-03
  Arms: PR Lotion Topical Solution
Other: Placebo Lotion — Placebo Topical Solution. Lotion will be created by the AMP Human Performance company and will include all ingredients similar to the PR Lotion product except for the exclusion of sodium bicarbonate.
  Arms: Placebo Lotion Topical Solution

SUMMARY:
The purpose of this research study is to evaluate the effects of a topical sodium bicarbonate lotion on physiological and psychological responses associated with hydration status and fluid balance in humans during passive heat stress. Currently, the ingestion of sodium has been an effective measure for improvements in fluid regulation and hydration status in humans. However, the investigators do not know its regulatory relationship with measurements of fluid balance when supplemented through the skin.

DETAILED DESCRIPTION:
Design This laboratory study is a randomized, counterbalanced, crossover design involving 20 participants (20 males) from the local community and university. This project will be conducted within the thermal physiology laboratory, complete with a climatic chamber (Cantrol, CES +13/+44) located within the Human Performance Laboratory (HPL) at the University of Connecticut. The investigators expect each interested individual will complete both phases included within the study design within a randomized, counterbalanced order.

Participant grouping orders will be randomly assigned by the project's lead student investigator (Jeb Struder). Each phase will be fairly similar in procedures completed; however, one phase will be completed with a trial that introduces a biomedical intervention (sodium bicarbonate topical lotion; PR group), while the other phase will be completed with a trial that introduces a placebo (PLA group) product similar to the biomedical intervention. Approximately 24 hours should pass between the completion of each session within a phase of the study. Additionally, approximately 3 days should pass between the completion of a phase and the initiation of the next phase (5th session completed).

Environmental Conditions Sessions I, II, and III of both counterbalanced groups (PR and PLA) will all be completed within thermoneutral conditions. Session IV of both counterbalanced groups (PR and PLA) will be conducted within the climatic chamber set to a climate with ambient temperature at approximately 33C (91.4F) and relative humidity at approximately 25%.

Baseline Assessments (PR/PLAI, PR/PLAII, PR/PLA III) Baseline visits should be completed over 3 consecutive days for the establishment of baseline measurements regarding the participant's body weight, dietary behaviors, and hydration status. Each assessment will be performed at the relatively same time of day (early to late morning) and will involve approximately 30 minutes spent within the laboratory space of the Human Performance Laboratory (HPL). All Baseline Assessment sessions will consist of fairly similar data collection procedures and will begin with the participant providing the completed 24-h dietary recall log, thirst perception scale, and filled urine jug to the administrating researcher. Additionally, the participant will be asked to provide a morning urine sample and nude body weight for the assessment of session-specific hydration status and Fluid Retention Index (FRI). Furthermore, once these tasks are completed, an HPL trained researcher will conduct a blood draw for the collection of approximately ½ teaspoon of blood. Each session will deviate slightly in additional tasks required for completion.

Day 1 (PR/PLAI): After the collection of a morning urine sample and nude body weight measurement, the participant's height (for additional anthropometrics) and resting blood pressure (for safety precautions) will be measured. Additionally, after the completion of the blood draw, the final task for this session will be the participant's familiarization to the Cognitive/Perceptual Battery tasks that you will be tested during Session 4 (PR/PLAIV).

Day 2 (PR/PLAII): After the collection of a morning urine sample and nude body weight measurement, the participant will be asked to rest within a comfortable position for approximately 10-15 minutes for the measurement of their resting heart rate.

Day 3 (PR/PLAIII): After the collection of a morning urine sample and nude body weight measurement, the participant will have their body fat percentage measured via handheld Lange Skinfold Calipers.

Intervention Trial (PR/PLAIV) Pre-Testing Procedures Prior to completing all Intervention Trial visits, participants will be asked to drink 500 mL of water before going to bed and an additional 500 mL of water upon waking to ensure proper hydration. If morning sample urine USG is ≤1.020, participants will be cleared to participate. If the participant arrives with a urine USG between 1.020 and 1.025, the subject will be asked to drink an additional 500 mL of water prior to entering the chamber to ensure proper hydration status. If participants arrive at the lab with a urine USG >1.025, the visit will be rescheduled for the following day. In addition to completing a morning urine spot sample, participants will be asked to complete a nude body mass measurement as well as provide their completed thirst perception scale, dietary recall log, and urine jug. Furthermore, using the urine and nude body weight measurements collected, the session-specific FRI will be assessed. Afterwards, the participant will be provided a standardized breakfast. Once the participant has indicated they are finished with their meal, resting blood pressure measurements will be conducted. Once all measurements have been completed, participants will have a venous cannula inserted by an HPL trained research team member. Finally, prior to entering the environmental chamber, participants will be instructed to privately insert the rectal thermometer 10-15 cm beyond the anal sphincter in addition to completing an additional nude body mass measurement and being fitted with a heart rate strap by the administrating research team.

Data Collection - Initial 120-minutes Upon the completion of participant arrival procedures, participants will then be permitted to enter the environmental chamber (~33C [91.4F], ~25% relative humidity) where they will be instructed to sit down and begin a 30-minute period of environmental equilibration. Once this period has been initiated the participant will be asked to complete their baseline measurements in regard to the Cognitive/Perceptual Battery. After the equilibration period has been completed, the participant will have their resting blood pressure measured, provide a baseline blood sample (~11 mL), and then provide both a urine sample and nude body weight measurement. Once all of these tasks have been completed, the participant will be provided approximately 50 g of the topical lotion (i.e. PR Lotion or Placebo) to apply to their upper body. Afterwards, blood samples (~3 mL) will be collected approximately 15- and 30-minutes post-lotion application. Furthermore, the hyperhydration protocol will be initiated at the 30-minute post-lotion application time point. During this time period, the first of 4 fluid boluses will be provided to the participant for consumption with instructions to consume all fluids provided within the allotted 15-minute time period before the provision of their next fluid bolus. Additionally, before the 3rd fluid bolus has been provided for consumption (identified as time point -30 min in Figure 4), another blood sample (~11 mL) will be completed before completing the rest of the hyperhydration protocol.

Hyperhydration Protocol To induce hyperhydration, participants will drink a total fluid volume of approximately 25 mL/kg of fat free mass (FFM) of water. These solutions will be pre-measured and provided within four enclosed water bottles for consumption at a rate of approximately 6.5 mL/kg FFM about every 15 minutes within a duration of approximately 60 minutes.

Topical Solution Procedures Approximately 50 grams of the topical solution will be pre-measured into 2 separate plastic bags and provided to the participant for application. Participants will be instructed to apply the solution primarily to areas of their upper extremities which will include an identified area from the wrist up to the clavicular area of the shoulder in addition to their chest, neck, upper back, midsection, and lower back if enough solution is available. Application will be considered complete when the solution has been transmitted to the skin in a fashion to where no residue from the lotion is visible by researchers from the skin of the participant.

Data Collection - 3-hour Protocol Collection of Blood Samples Aside from the baseline blood sample collected around the -90-minute time point, an initial blood sample will occur at time point 0 min, where approximately 11 mL of blood will be collected via the inserted cannula. Similar blood samples will be collected at time intervals of approximately 60-minutes up to the completion of the data collection protocol, occurring around the 180-minute mark (approximately 3-hours). In total, approximately 72 mL of blood will be collected during the Intervention Trial, which is less than ¼ of the amount of blood collected during a blood donation.

Collection of Urine Samples and Body Weight Measurements For the collection of all urine spot samples, researchers will provide a clean cup and top to seal the capsule. Participants will be asked to provide a sample regardless of urgency to urinate at specific time points during the trial. If the participant is unable to provide a sample at the time point requested, no protocol deviation will be considered as the lack in sample provided will still be used towards the completion of data analysis. Furthermore, if the participant must provide a urine sample without being requested by a research team member, any urine expelled will be added to the amount collected (if any) during the next urine sample collection time point. Additionally, participants will be instructed to complete a measurement of nude body weight completed before the provision of a urine sample. Both the collection of urine samples and measurement of body weight will be completed within the privacy of a bathroom. Aside from the baseline measurement completed around the -90-minute time point, the initial urine sample collection and body weight measurement for the intervention (i.e. PR Lotion or Placebo) will approximately occur at time point 0-minutes and supplementary urine collection and body weight measurement will be completed in 30-minute intervals up to the end of the data collection period, occurring around the 180-minute mark (approximately 3-hours).

Completion of Cognitive/Perceptual Battery Aside from the baseline Cognitive/Perceptual Battery completed around the -115-minute time point, the initial Cognitive/Perceptual Battery will be completed at time point 0-minutes. Completion of supplemental Cognitive/Perceptual Batteries will be continually measured within a 60-minute time interval from time point 0-minutes until the completion of data collection which will coincide with the 180-minute time point (approximately 3-hours).

ELIGIBILITY:
Inclusion Criteria:

1. Males within the age range of 18-35 years old.
2. Individuals who are classified as recreationally active individuals: physical activity performed ≥3 days per week with sessions lasting ≥30 minutes in duration.
3. Individuals who have been medically cleared for participation in this study by the medical safety monitor.

Exclusion Criteria:

1. Cannot understand English (written and/or verbally communicated).
2. Hearing impaired to where verbal communications cannot be understood and/or followed safely.
3. Individuals who self-report history of complications with psychological disorders or chronic illness (eating disorders, cardiovascular, kidney, liver, metabolic, neuromuscular, pulmonary, and/or sickle cell disease).
4. Individuals who have chronic health problems that may affect the participant's ability to thermoregulate or sweat normally.
5. Individuals who have a history of exertional heat illness within the past 3 years.
6. Individuals who are taking any prescription or non-prescription medication(s) that may specifically impact cardiometabolic, pulmonary, renal, and/or thermoregulatory function (i.e. amphetamines, antihypertensives, anticholinergics, acetaminophen, NSAIDs, aspirin, and water pills).
7. Individuals who have consumed more than (>3,500 mg) or less than (<2,300 mg) the average amount of sodium consumed per day at time of testing.
8. Individuals who have consumed more than (>1.8L) or less than (<0.8L) the average amount of fluids consumed per day at time of testing.
9. Individuals classified as hypertensive while at rest (SBP: ≥140 mmHg and/or DBP: ≥90 mmHg; will be measured during first visit).
10. Individuals who have not abstained from use of supplements that may affect/enhance hydration status (i.e. creatine, sodium bicarbonate, potassium, magnesium, dandelion, vitamin B6, other natural diuretics) at time of testing.
11. Individuals who report they are suffering from a fever or current illness at time of testing.
12. Individuals who are suffering from a current musculoskeletal injury that limits the participant's ability to walk, stand, and/or sit upright in a chair for long periods of time.
13. Individuals who have an active lesion at the location of topical solution application.
14. Individuals how are allergic/sensitive to ingredients within the study-specific Topical Lotions: (Menthol [0.5%], sodium bicarbonate (baking soda), water, isopropyl palmitate, lecithin, poloxamer 407, cetyl alcohol, propylene glycol, denatured alcohol, benzyl alcohol, polyglyceryl-4 laurate, sodium hydroxide, sodium lauryl sulfate, sorbic acid, and fragrance).
15. Individuals who are allergic/sensitive to iodine, water-based ultrasound solution, and/or medical tape.
16. Individuals who have experienced any recent major life events (i.e. death in family, divorce, wedding) in the previous 6 months.
17. Individuals who have donated blood within the previous month.
18. Individuals who have an implanted pacemaker or internal defibrillator.
19. Individuals who use tobacco products (including smoking cessation products).

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
Fluid Retention - Change in Expelled Urine Volume | Hydration Baseline Day 1
  Assessment of fluid retention via collection of urine volume
Fluid Retention - Change in Expelled Urine Volume | Hydration Baseline Day 2
  Assessment of fluid retention via collection of urine volume
Fluid Retention - Change in Expelled Urine Volume | Hydration Baseline Day 3
  Assessment of fluid retention via collection of urine volume
Fluid Retention - Change in Expelled Urine Volume | Intervention Trial (Day 4) at the -90 minute mark.
  Assessment of fluid retention via collection of urine volume
Fluid Retention - Change in Expelled Urine Volume | Intervention Trial (Day 4) at the 0 minute mark.
  Assessment of fluid retention via collection of urine volume
Fluid Retention - Change in Expelled Urine Volume | Intervention Trial (Day 4) at the 30 minute mark.
  Assessment of fluid retention via collection of urine volume
Fluid Retention - Change in Expelled Urine Volume | Intervention Trial (Day 4) at the 60 minute mark.
  Assessment of fluid retention via collection of urine volume
Fluid Retention - Change in Expelled Urine Volume | Intervention Trial (Day 4) at the 90 minute mark.
  Assessment of fluid retention via collection of urine volume
Fluid Retention - Change in Expelled Urine Volume | Intervention Trial (Day 4) at the 120 minute mark.
  Assessment of fluid retention via collection of urine volume
Fluid Retention - Change in Expelled Urine Volume | Intervention Trial (Day 4) at the 180 minute mark.
  Assessment of fluid retention via collection of urine volume
Kidney Function - Change in Aldosterone Response | Hydration Baseline Day 1
  Assessment of kidney function in regards to fluid retention via assessment of blood biomarkers associated with kidney function
Kidney Function - Change in Aldosterone Response | Hydration Baseline Day 2
  Assessment of kidney function in regards to fluid retention via assessment of blood biomarkers associated with kidney function
Kidney Function - Change in Aldosterone Response | Hydration Baseline Day 3
  Assessment of kidney function in regards to fluid retention via assessment of blood biomarkers associated with kidney function
Kidney Function - Change in Aldosterone Response | Intervention Trial (Day 4) at the -90 minute mark.
  Assessment of kidney function in regards to fluid retention via assessment of blood biomarkers associated with kidney function
Kidney Function - Change in Aldosterone Response | Intervention Trial (Day 4) at the -30 minute mark.
  Assessment of kidney function in regards to fluid retention via assessment of blood biomarkers associated with kidney function
Kidney Function - Change in Aldosterone Response | Intervention Trial (Day 4) at the 0 minute mark.
  Assessment of kidney function in regards to fluid retention via assessment of blood biomarkers associated with kidney function
Kidney Function - Change in Aldosterone Response | Intervention Trial (Day 4) at the 60 minute mark.
  Assessment of kidney function in regards to fluid retention via assessment of blood biomarkers associated with kidney function
Kidney Function - Change in Aldosterone Response | Intervention Trial (Day 4) at the 120 minute mark.
  Assessment of kidney function in regards to fluid retention via assessment of blood biomarkers associated with kidney function
Kidney Function - Change in Aldosterone Response | Intervention Trial (Day 4) at the 180 minute mark.
  Assessment of kidney function in regards to fluid retention via assessment of blood biomarkers associated with kidney function
Kidney Function - Change in Copeptin Response | Hydration Baseline Day 1
  Assessment of kidney function in regards to fluid retention via assessment of blood biomarkers associated with kidney function
Kidney Function - Change in Copeptin Response | Hydration Baseline Day 2
  Assessment of kidney function in regards to fluid retention via assessment of blood biomarkers associated with kidney function
Kidney Function - Change in Copeptin Response | Hydration Baseline Day 3
  Assessment of kidney function in regards to fluid retention via assessment of blood biomarkers associated with kidney function
Kidney Function - Change in Copeptin Response | Intervention Trial (Day 4) at the -90 minute mark.
  Assessment of kidney function in regards to fluid retention via assessment of blood biomarkers associated with kidney function
Kidney Function - Change in Copeptin Response | Intervention Trial (Day 4) at the -30 minute mark.
  Assessment of kidney function in regards to fluid retention via assessment of blood biomarkers associated with kidney function
Kidney Function - Change in Copeptin Response | Intervention Trial (Day 4) at the 0 minute mark.
  Assessment of kidney function in regards to fluid retention via assessment of blood biomarkers associated with kidney function
Kidney Function - Change in Copeptin Response | Intervention Trial (Day 4) at the 60 minute mark.
  Assessment of kidney function in regards to fluid retention via assessment of blood biomarkers associated with kidney function
Kidney Function - Change in Copeptin Response | Intervention Trial (Day 4) at the 120 minute mark.
  Assessment of kidney function in regards to fluid retention via assessment of blood biomarkers associated with kidney function
Kidney Function - Change in Copeptin Response | Intervention Trial (Day 4) at the 180 minute mark.
  Assessment of kidney function in regards to fluid retention via assessment of blood biomarkers associated with kidney function
Kidney Function - Change in Creatinine Response | Hydration Baseline Day 1
  Assessment of kidney function in regards to fluid retention via assessment of urine biomarkers associated with kidney function
Kidney Function - Change in Creatinine Response | Hydration Baseline Day 2
  Assessment of kidney function in regards to fluid retention via assessment of urine biomarkers associated with kidney function
Kidney Function - Change in Creatinine Response | Hydration Baseline Day 3
  Assessment of kidney function in regards to fluid retention via assessment of urine biomarkers associated with kidney function
Kidney Function - Change in Creatinine Response | Intervention Trial (Day 4) at the -90 minute mark.
  Assessment of kidney function in regards to fluid retention via assessment of urine biomarkers associated with kidney function
Kidney Function - Change in Creatinine Response | Intervention Trial (Day 4) at the 0 minute mark.
  Assessment of kidney function in regards to fluid retention via assessment of urine biomarkers associated with kidney function
Kidney Function - Change in Creatinine Response | Intervention Trial (Day 4) at the 60 minute mark.
  Assessment of kidney function in regards to fluid retention via assessment of urine biomarkers associated with kidney function
Kidney Function - Change in Creatinine Response | Intervention Trial (Day 4) at the 120 minute mark.
  Assessment of kidney function in regards to fluid retention via assessment of urine biomarkers associated with kidney function
Kidney Function - Change in Creatinine Response | Intervention Trial (Day 4) at the 180 minute mark.
  Assessment of kidney function in regards to fluid retention via assessment of urine biomarkers associated with kidney function
Change in Whole Blood Sodium Levels | Hydration Baseline Day 1
  Assessment of fluid retention via whole blood sodium (electrolyte levels) through blood biomarkers
Change in Whole Blood Sodium Levels | Hydration Baseline Day 2
  Assessment of fluid retention via whole blood sodium (electrolyte levels) through blood biomarkers
Change in Whole Blood Sodium Levels | Hydration Baseline Day 3
  Assessment of fluid retention via whole blood sodium (electrolyte levels) through blood biomarkers
Change in Whole Blood Sodium Levels | Intervention Trial (Day 4) at the -90 minute mark.
  Assessment of fluid retention via whole blood sodium (electrolyte levels) through blood biomarkers
Change in Whole Blood Sodium Levels | Intervention Trial (Day 4) at the -75 minute mark.
  Assessment of fluid retention via whole blood sodium (electrolyte levels) through blood biomarkers
Change in Whole Blood Sodium Levels | Intervention Trial (Day 4) at the -60 minute mark.
  Assessment of fluid retention via whole blood sodium (electrolyte levels) through blood biomarkers
Change in Whole Blood Sodium Levels | Intervention Trial (Day 4) at the -30 minute mark.
  Assessment of fluid retention via whole blood sodium (electrolyte levels) through blood biomarkers
Change in Whole Blood Sodium Levels | Intervention Trial (Day 4) at the 0 minute mark.
  Assessment of fluid retention via whole blood sodium (electrolyte levels) through blood biomarkers
Change in Whole Blood Sodium Levels | Intervention Trial (Day 4) at the 60 minute mark.
  Assessment of fluid retention via whole blood sodium (electrolyte levels) through blood biomarkers
Change in Whole Blood Sodium Levels | Intervention Trial (Day 4) at the 120 minute mark.
  Assessment of fluid retention via whole blood sodium (electrolyte levels) through blood biomarkers
Change in Whole Blood Sodium Levels | Intervention Trial (Day 4) at the 180 minute mark.
  Assessment of fluid retention via whole blood sodium (electrolyte levels) through blood biomarkers
Change in Whole Blood Potassium Levels | Hydration Baseline Day 1
  Assessment of fluid retention via whole blood potassium (electrolyte levels) through blood biomarkers
Change in Whole Blood Potassium Levels | Hydration Baseline Day 2
  Assessment of fluid retention via whole blood potassium (electrolyte levels) through blood biomarkers
Change in Whole Blood Potassium Levels | Hydration Baseline Day 3
  Assessment of fluid retention via whole blood potassium (electrolyte levels) through blood biomarkers
Change in Whole Blood Potassium Levels | Intervention Trial (Day 4) at the -90 minute mark.
  Assessment of fluid retention via whole blood potassium (electrolyte levels) through blood biomarkers
Change in Whole Blood Potassium Levels | Intervention Trial (Day 4) at the -75 minute mark.
  Assessment of fluid retention via whole blood potassium (electrolyte levels) through blood biomarkers
Change in Whole Blood Potassium Levels | Intervention Trial (Day 4) at the -60 minute mark.
  Assessment of fluid retention via whole blood potassium (electrolyte levels) through blood biomarkers
Change in Whole Blood Potassium Levels | Intervention Trial (Day 4) at the -30 minute mark.
  Assessment of fluid retention via whole blood potassium (electrolyte levels) through blood biomarkers
Change in Whole Blood Potassium Levels | Intervention Trial (Day 4) at the 0 minute mark.
  Assessment of fluid retention via whole blood potassium (electrolyte levels) through blood biomarkers
Change in Whole Blood Potassium Levels | Intervention Trial (Day 4) at the 60 minute mark.
  Assessment of fluid retention via whole blood potassium (electrolyte levels) through blood biomarkers
Change in Whole Blood Potassium Levels | Intervention Trial (Day 4) at the 120 minute mark.
  Assessment of fluid retention via whole blood potassium (electrolyte levels) through blood biomarkers
Change in Whole Blood Potassium Levels | Intervention Trial (Day 4) at the 180 minute mark.
  Assessment of fluid retention via whole blood potassium (electrolyte levels) through blood biomarkers
Change in Whole Blood Chloride Levels | Hydration Baseline Day 1
  Assessment of fluid retention via whole blood chloride (electrolyte levels) through blood biomarkers
Change in Whole Blood Chloride Levels | Hydration Baseline Day 2
  Assessment of fluid retention via whole blood chloride (electrolyte levels) through blood biomarkers
Change in Whole Blood Chloride Levels | Hydration Baseline Day 3
  Assessment of fluid retention via whole blood chloride (electrolyte levels) through blood biomarkers
Change in Whole Blood Chloride Levels | Intervention Trial (Day 4) at the -90 minute mark.
  Assessment of fluid retention via whole blood chloride (electrolyte levels) through blood biomarkers
Change in Whole Blood Chloride Levels | Intervention Trial (Day 4) at the -75 minute mark.
  Assessment of fluid retention via whole blood chloride (electrolyte levels) through blood biomarkers
Change in Whole Blood Chloride Levels | Intervention Trial (Day 4) at the -60 minute mark.
  Assessment of fluid retention via whole blood chloride (electrolyte levels) through blood biomarkers
Change in Whole Blood Chloride Levels | Intervention Trial (Day 4) at the -30 minute mark.
  Assessment of fluid retention via whole blood chloride (electrolyte levels) through blood biomarkers
Change in Whole Blood Chloride Levels | Intervention Trial (Day 4) at the 0 minute mark.
  Assessment of fluid retention via whole blood chloride (electrolyte levels) through blood biomarkers
Change in Whole Blood Chloride Levels | Intervention Trial (Day 4) at the 60 minute mark.
  Assessment of fluid retention via whole blood chloride (electrolyte levels) through blood biomarkers
Change in Whole Blood Chloride Levels | Intervention Trial (Day 4) at the 120 minute mark.
  Assessment of fluid retention via whole blood chloride (electrolyte levels) through blood biomarkers
Change in Whole Blood Chloride Levels | Intervention Trial (Day 4) at the 180 minute mark.
  Assessment of fluid retention via whole blood chloride (electrolyte levels) through blood biomarkers

SECONDARY OUTCOMES:
Fluid Retention - Change in Whole Blood Hematocrit Levels | Hydration Baseline 1
  Assessment of plasma volume shifts which may indicate fluid retention via assessment of changes in hematocrit levels
Fluid Retention - Change in Whole Blood Hematocrit Levels | Hydration Baseline 2
  Assessment of plasma volume shifts which may indicate fluid retention via assessment of changes in hematocrit levels
Fluid Retention - Change in Whole Blood Hematocrit Levels | Hydration Baseline 3
  Assessment of plasma volume shifts which may indicate fluid retention via assessment of changes in hematocrit levels
Fluid Retention - Change in Whole Blood Hematocrit Levels | Intervention Trial (Day 4) at the -90 minute mark.
  Assessment of plasma volume shifts which may indicate fluid retention via assessment of changes in hematocrit levels
Fluid Retention - Change in Whole Blood Hematocrit Levels | Intervention Trial (Day 4) at the -75 minute mark.
  Assessment of plasma volume shifts which may indicate fluid retention via assessment of changes in hematocrit levels
Fluid Retention - Change in Whole Blood Hematocrit Levels | Intervention Trial (Day 4) at the -60 minute mark.
  Assessment of plasma volume shifts which may indicate fluid retention via assessment of changes in hematocrit levels
Fluid Retention - Change in Whole Blood Hematocrit Levels | Intervention Trial (Day 4) at the -30 minute mark.
  Assessment of plasma volume shifts which may indicate fluid retention via assessment of changes in hematocrit levels
Fluid Retention - Change in Whole Blood Hematocrit Levels | Intervention Trial (Day 4) at the 0 minute mark.
  Assessment of plasma volume shifts which may indicate fluid retention via assessment of changes in hematocrit levels
Fluid Retention - Change in Whole Blood Hematocrit Levels | Intervention Trial (Day 4) at the 60 minute mark.
  Assessment of plasma volume shifts which may indicate fluid retention via assessment of changes in hematocrit levels
Fluid Retention - Change in Whole Blood Hematocrit Levels | Intervention Trial (Day 4) at the 120 minute mark.
  Assessment of plasma volume shifts which may indicate fluid retention via assessment of changes in hematocrit levels
Fluid Retention - Change in Whole Blood Hematocrit Levels | Intervention Trial (Day 4) at the 180 minute mark.
  Assessment of plasma volume shifts which may indicate fluid retention via assessment of changes in hematocrit levels
Fluid Retention - Change in Whole Blood Hemoglobin Levels | Hydration Baseline Day 1
  Assessment of plasma volume shifts which may indicate fluid retention via assessment of changes in hemoglobin levels
Fluid Retention - Change in Whole Blood Hemoglobin Levels | Hydration Baseline Day 2
  Assessment of plasma volume shifts which may indicate fluid retention via assessment of changes in hemoglobin levels
Fluid Retention - Change in Whole Blood Hemoglobin Levels | Hydration Baseline Day 3
  Assessment of plasma volume shifts which may indicate fluid retention via assessment of changes in hemoglobin levels
Fluid Retention - Change in Whole Blood Hemoglobin Levels | Intervention Trial (Day 4) at the -90 minute mark.
  Assessment of plasma volume shifts which may indicate fluid retention via assessment of changes in hemoglobin levels
Fluid Retention - Change in Whole Blood Hemoglobin Levels | Intervention Trial (Day 4) at the -75 minute mark.
  Assessment of plasma volume shifts which may indicate fluid retention via assessment of changes in hemoglobin levels
Fluid Retention - Change in Whole Blood Hemoglobin Levels | Intervention Trial (Day 4) at the -60 minute mark.
  Assessment of plasma volume shifts which may indicate fluid retention via assessment of changes in hemoglobin levels
Fluid Retention - Change in Whole Blood Hemoglobin Levels | Intervention Trial (Day 4) at the -30 minute mark.
  Assessment of plasma volume shifts which may indicate fluid retention via assessment of changes in hemoglobin levels
Fluid Retention - Change in Whole Blood Hemoglobin Levels | Intervention Trial (Day 4) at the 0 minute mark.
  Assessment of plasma volume shifts which may indicate fluid retention via assessment of changes in hemoglobin levels
Fluid Retention - Change in Whole Blood Hemoglobin Levels | Intervention Trial (Day 4) at the 60 minute mark.
  Assessment of plasma volume shifts which may indicate fluid retention via assessment of changes in hemoglobin levels
Fluid Retention - Change in Whole Blood Hemoglobin Levels | Intervention Trial (Day 4) at the 120 minute mark.
  Assessment of plasma volume shifts which may indicate fluid retention via assessment of changes in hemoglobin levels
Fluid Retention - Change in Whole Blood Hemoglobin Levels | Intervention Trial (Day 4) at the 180 minute mark.
  Assessment of plasma volume shifts which may indicate fluid retention via assessment of changes in hemoglobin levels
Fluid Retention - Change in Plasma Osmolality Shifts | Hydration Baseline Day 1
  Assessment of fluid retention via changes in plasma osmolality
Fluid Retention - Change in Plasma Osmolality Shifts | Hydration Baseline Day 2
  Assessment of fluid retention via changes in plasma osmolality
Fluid Retention - Change in Plasma Osmolality Shifts | Hydration Baseline Day 3
  Assessment of fluid retention via changes in plasma osmolality
Fluid Retention - Change in Plasma Osmolality Shifts | Intervention Trial (Day 4) at the -90 minute mark.
  Assessment of fluid retention via changes in plasma osmolality
Fluid Retention - Change in Plasma Osmolality Shifts | Intervention Trial (Day 4) at the -75 minute mark.
  Assessment of fluid retention via changes in plasma osmolality
Fluid Retention - Change in Plasma Osmolality Shifts | Intervention Trial (Day 4) at the -60 minute mark.
  Assessment of fluid retention via changes in plasma osmolality
Fluid Retention - Change in Plasma Osmolality Shifts | Intervention Trial (Day 4) at the -30 minute mark.
  Assessment of fluid retention via changes in plasma osmolality
Fluid Retention - Change in Plasma Osmolality Shifts | Intervention Trial (Day 4) at the 0 minute mark.
  Assessment of fluid retention via changes in plasma osmolality
Fluid Retention - Change in Plasma Osmolality Shifts | Intervention Trial (Day 4) at the 60 minute mark.
  Assessment of fluid retention via changes in plasma osmolality
Fluid Retention - Change in Plasma Osmolality Shifts | Intervention Trial (Day 4) at the 120 minute mark.
  Assessment of fluid retention via changes in plasma osmolality
Fluid Retention - Change in Plasma Osmolality Shifts | Intervention Trial (Day 4) at the 180 minute mark.
  Assessment of fluid retention via changes in plasma osmolality
Kidney Function - Change in Urine Color | Hydration Baseline Day 1
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Color | Hydration Baseline Day 2
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Color | Hydration Baseline Day 3
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Color | Intervention Trial (Day 4) at the -90 minute mark.
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Color | Intervention Trial (Day 4) at the 0 minute mark.
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Color | Intervention Trial (Day 4) at the 30 minute mark.
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Color | Intervention Trial (Day 4) at the 60 minute mark.
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Color | Intervention Trial (Day 4) at the 90 minute mark.
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Color | Intervention Trial (Day 4) at the 120 minute mark.
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Color | Intervention Trial (Day 4) at the 150 minute mark.
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Color | Intervention Trial (Day 4) at the 180 minute mark.
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Specific Gravity | Hydration Baseline Day 1
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Specific Gravity | Hydration Baseline Day 2
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Specific Gravity | Hydration Baseline Day 3
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Specific Gravity | Intervention Trial (Day 4) at the -90 minute mark.
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Specific Gravity | Intervention Trial (Day 4) at the 0 minute mark.
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Specific Gravity | Intervention Trial (Day 4) at the 30 minute mark.
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Specific Gravity | Intervention Trial (Day 4) at the 60 minute mark.
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Specific Gravity | Intervention Trial (Day 4) at the 90 minute mark.
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Specific Gravity | Intervention Trial (Day 4) at the 120 minute mark.
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Specific Gravity | Intervention Trial (Day 4) at the 150 minute mark.
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Specific Gravity | Intervention Trial (Day 4) at the 180 minute mark.
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Osmolality | Hydration Baseline Day 1
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Osmolality | Hydration Baseline Day 2
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Osmolality | Hydration Baseline Day 3
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Osmolality | Intervention Trial (Day 4) at the -90 minute mark.
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Osmolality | Intervention Trial (Day 4) at the 0 minute mark.
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Osmolality | Intervention Trial (Day 4) at the 30 minute mark.
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Osmolality | Intervention Trial (Day 4) at the 60 minute mark.
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Osmolality | Intervention Trial (Day 4) at the 90 minute mark.
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Osmolality | Intervention Trial (Day 4) at the 120 minute mark.
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Osmolality | Intervention Trial (Day 4) at the 150 minute mark.
  Assessment of kidney function via urine biomarkers collected during data procedures.
Kidney Function - Change in Urine Osmolality | Intervention Trial (Day 4) at the 180 minute mark.
  Assessment of kidney function via urine biomarkers collected during data procedures.
Cardiovascular Function - Change in Blood Pressure | Hydration Baseline Day 1
  Assessment of cardiovascular function via blood pressure changes during data collection procedures
Cardiovascular Function - Change in Blood Pressure | Intervention Trial (Day 4) at the -90 minute mark.
  Assessment of cardiovascular function via blood pressure changes during data collection procedures
Cardiovascular Function - Change in Blood Pressure | Intervention Trial (Day 4) at the 0 minute mark.
  Assessment of cardiovascular function via blood pressure changes during data collection procedures
Cardiovascular Function - Change in Blood Pressure | Intervention Trial (Day 4) at the 30 minute mark.
  Assessment of cardiovascular function via blood pressure changes during data collection procedures
Cardiovascular Function - Change in Blood Pressure | Intervention Trial (Day 4) at the 90 minute mark.
  Assessment of cardiovascular function via blood pressure changes during data collection procedures
Cardiovascular Function - Change in Blood Pressure | Intervention Trial (Day 4) at the 150 minute mark.
  Assessment of cardiovascular function via blood pressure changes during data collection procedures
Cardiovascular Function - Change in Heart Rate Variability | Hydration Baseline Day 2
  Assessment of cardiovascular function via heart rate variability changes during data collection procedures
Cardiovascular Function - Change in Heart Rate Variability | Intervention Trial (Day 4) at the -90 minute mark
  Assessment of cardiovascular function via heart rate variability changes during data collection procedures
Cardiovascular Function - Change in Heart Rate Variability | Intervention Trial (Day 4) at the 0 minute mark
  Assessment of cardiovascular function via heart rate variability changes during data collection procedures
Cardiovascular Function - Change in Heart Rate Variability | Intervention Trial (Day 4) at the 30 minute mark
  Assessment of cardiovascular function via heart rate variability changes during data collection procedures
Cardiovascular Function - Change in Heart Rate Variability | Intervention Trial (Day 4) at the 90 minute mark
  Assessment of cardiovascular function via heart rate variability changes during data collection procedures
Cardiovascular Function - Change in Heart Rate Variability | Intervention Trial (Day 4) at the 150 minute mark
  Assessment of cardiovascular function via heart rate variability changes during data collection procedures
Cardiovascular Function - Change in Resting Heart Rate | Intervention Trial (Day 4)
  Assessment of cardiovascular function via resting heart rate changes during data collection procedures
Cognitive Differences - Changes in Go/No Go Assessment | Intervention Trial (Day 4) at the -115 minute mark.
  This test will be used for the assessment of response inhibition. For completion of the test, the participant will be presented with two characters, "x" and "o", and will be expected to either respond as quickly as possible ("x") or not ("o") depending on the visual stimulus provided.
Cognitive Differences - Changes in Go/No Go Assessment | Intervention Trial (Day 4) at the 0 minute mark.
  This test will be used for the assessment of response inhibition. For completion of the test, the participant will be presented with two characters, "x" and "o", and will be expected to either respond as quickly as possible ("x") or not ("o") depending on the visual stimulus provided.
Cognitive Differences - Changes in Go/No Go Assessment | Intervention Trial (Day 4) at the 60 minute mark.
  This test will be used for the assessment of response inhibition. For completion of the test, the participant will be presented with two characters, "x" and "o", and will be expected to either respond as quickly as possible ("x") or not ("o") depending on the visual stimulus provided.
Cognitive Differences - Changes in Go/No Go Assessment | Intervention Trial (Day 4) at the 120 minute mark.
  This test will be used for the assessment of response inhibition. For completion of the test, the participant will be presented with two characters, "x" and "o", and will be expected to either respond as quickly as possible ("x") or not ("o") depending on the visual stimulus provided.
Cognitive Differences - Changes in Go/No Go Assessment | Intervention Trial (Day 4) at the 180 minute mark.
  This test will be used for the assessment of response inhibition. For completion of the test, the participant will be presented with two characters, "x" and "o", and will be expected to either respond as quickly as possible ("x") or not ("o") depending on the visual stimulus provided.
Cognitive Differences - Changes in 2 Choice Reaction Time | Intervention Trial (Day 4) at the -115 minute mark.
  This test will be used for the assessment of attention and processing speed when presented with the opportunity to make a simple choice. The test will include a "*" or "o" which will be presented on the computer screen display. The participant will be instructed to respond as quickly as possible by pressing the designated button for each stimulus as it appears on the screen.
Cognitive Differences - Changes in 2 Choice Reaction Time | Intervention Trial (Day 4) at the 0 minute mark.
  This test will be used for the assessment of attention and processing speed when presented with the opportunity to make a simple choice. The test will include a "*" or "o" which will be presented on the computer screen display. The participant will be instructed to respond as quickly as possible by pressing the designated button for each stimulus as it appears on the screen.
Cognitive Differences - Changes in 2 Choice Reaction Time | Intervention Trial (Day 4) at the 60 minute mark.
  This test will be used for the assessment of attention and processing speed when presented with the opportunity to make a simple choice. The test will include a "*" or "o" which will be presented on the computer screen display. The participant will be instructed to respond as quickly as possible by pressing the designated button for each stimulus as it appears on the screen.
Cognitive Differences - Changes in 2 Choice Reaction Time | Intervention Trial (Day 4) at the 120 minute mark.
  This test will be used for the assessment of attention and processing speed when presented with the opportunity to make a simple choice. The test will include a "*" or "o" which will be presented on the computer screen display. The participant will be instructed to respond as quickly as possible by pressing the designated button for each stimulus as it appears on the screen.
Cognitive Differences - Changes in 2 Choice Reaction Time | Intervention Trial (Day 4) at the 180 minute mark.
  This test will be used for the assessment of attention and processing speed when presented with the opportunity to make a simple choice. The test will include a "*" or "o" which will be presented on the computer screen display. The participant will be instructed to respond as quickly as possible by pressing the designated button for each stimulus as it appears on the screen.
Cognitive Differences - Changes in Procedural Reaction Time | Intervention Trial (Day 4) at the -115 minute mark.
  This test will be associated with the comprehension of a simple set of rules provided to participants during testing completion and will be used for the assessment of reaction time and processing efficiency. Participants will be presented with a number constructed using a large dot matrix on the computer display. Participants will be tasked with pressing a button correctly designated towards the identification of a "low" number or "high" number.
Cognitive Differences - Changes in Procedural Reaction Time | Intervention Trial (Day 4) at the 0 minute mark.
  This test will be associated with the comprehension of a simple set of rules provided to participants during testing completion and will be used for the assessment of reaction time and processing efficiency. Participants will be presented with a number constructed using a large dot matrix on the computer display. Participants will be tasked with pressing a button correctly designated towards the identification of a "low" number or "high" number.
Cognitive Differences - Changes in Procedural Reaction Time | Intervention Trial (Day 4) at the 60 minute mark.
  This test will be associated with the comprehension of a simple set of rules provided to participants during testing completion and will be used for the assessment of reaction time and processing efficiency. Participants will be presented with a number constructed using a large dot matrix on the computer display. Participants will be tasked with pressing a button correctly designated towards the identification of a "low" number or "high" number.
Cognitive Differences - Changes in Procedural Reaction Time | Intervention Trial (Day 4) at the 120 minute mark.
  This test will be associated with the comprehension of a simple set of rules provided to participants during testing completion and will be used for the assessment of reaction time and processing efficiency. Participants will be presented with a number constructed using a large dot matrix on the computer display. Participants will be tasked with pressing a button correctly designated towards the identification of a "low" number or "high" number.
Cognitive Differences - Changes in Procedural Reaction Time | Intervention Trial (Day 4) at the 180 minute mark.
  This test will be associated with the comprehension of a simple set of rules provided to participants during testing completion and will be used for the assessment of reaction time and processing efficiency. Participants will be presented with a number constructed using a large dot matrix on the computer display. Participants will be tasked with pressing a button correctly designated towards the identification of a "low" number or "high" number.
Cognitive Differences - Changes in Stroop Test | Intervention Trial (Day 4) at the -115 minute mark.
  This test will be used for the assessment of processing speed, selective attention, interference, and executive functioning skills by correctly identifying either the word- or color-based stimuli presented on the computer screen.
Cognitive Differences - Changes in Stroop Test | Intervention Trial (Day 4) at the 0 minute mark.
  This test will be used for the assessment of processing speed, selective attention, interference, and executive functioning skills by correctly identifying either the word- or color-based stimuli presented on the computer screen.
Cognitive Differences - Changes in Stroop Test | Intervention Trial (Day 4) at the 60 minute mark.
  This test will be used for the assessment of processing speed, selective attention, interference, and executive functioning skills by correctly identifying either the word- or color-based stimuli presented on the computer screen.
Cognitive Differences - Changes in Stroop Test | Intervention Trial (Day 4) at the 120 minute mark.
  This test will be used for the assessment of processing speed, selective attention, interference, and executive functioning skills by correctly identifying either the word- or color-based stimuli presented on the computer screen.
Cognitive Differences - Changes in Stroop Test | Intervention Trial (Day 4) at the 180 minute mark.
  This test will be used for the assessment of processing speed, selective attention, interference, and executive functioning skills by correctly identifying either the word- or color-based stimuli presented on the computer screen.
Perceptual Differences - Changes in Environmental Symptoms Questionnaire | Intervention Trial (Day 4) at the -115 minute mark.
  A modified version of the 68-item questionnaire will be administered. This is a test to monitor for symptoms of exertional heat illness (i.e. headache, dizziness, nausea, thirst, cramps, etc.) and will be administered during all sessions performed within environmental conditions.
Perceptual Differences - Changes in Environmental Symptoms Questionnaire | Intervention Trial (Day 4) at the 0 minute mark.
  A modified version of the 68-item questionnaire will be administered. This is a test to monitor for symptoms of exertional heat illness (i.e. headache, dizziness, nausea, thirst, cramps, etc.) and will be administered during all sessions performed within environmental conditions.
Perceptual Differences - Changes in Environmental Symptoms Questionnaire | Intervention Trial (Day 4) at the 60 minute mark.
  A modified version of the 68-item questionnaire will be administered. This is a test to monitor for symptoms of exertional heat illness (i.e. headache, dizziness, nausea, thirst, cramps, etc.) and will be administered during all sessions performed within environmental conditions.
Perceptual Differences - Changes in Environmental Symptoms Questionnaire | Intervention Trial (Day 4) at the 120 minute mark.
  A modified version of the 68-item questionnaire will be administered. This is a test to monitor for symptoms of exertional heat illness (i.e. headache, dizziness, nausea, thirst, cramps, etc.) and will be administered during all sessions performed within environmental conditions.
Perceptual Differences - Changes in Environmental Symptoms Questionnaire | Intervention Trial (Day 4) at the 180 minute mark.
  A modified version of the 68-item questionnaire will be administered. This is a test to monitor for symptoms of exertional heat illness (i.e. headache, dizziness, nausea, thirst, cramps, etc.) and will be administered during all sessions performed within environmental conditions.
Perceptual Differences - Changes in Fatigue Scale | Intervention Trial (Day 4) at the -115 minute mark.
  This scale has been associated with good face validity and high levels of convergent validity during exhaustive exercise.16 It consists of an eleven-point (0-10) Likert Scale with verbal anchors of 0, "No Fatigue At All", 1, "Very Small Amount of Fatigue", 2, "Small Amount of Fatigue", 3, "Moderate Fatigue", 4, "Somewhat Fatigued", 5, "Fatigued", 7, "Very Fatigued", 9, "Extremely Fatigued", and 10, "Completely Fatigued"
Perceptual Differences - Changes in Fatigue Scale | Intervention Trial (Day 4) at the 0 minute mark.
  This scale has been associated with good face validity and high levels of convergent validity during exhaustive exercise.16 It consists of an eleven-point (0-10) Likert Scale with verbal anchors of 0, "No Fatigue At All", 1, "Very Small Amount of Fatigue", 2, "Small Amount of Fatigue", 3, "Moderate Fatigue", 4, "Somewhat Fatigued", 5, "Fatigued", 7, "Very Fatigued", 9, "Extremely Fatigued", and 10, "Completely Fatigued"
Perceptual Differences - Changes in Fatigue Scale | Intervention Trial (Day 4) at the 60 minute mark.
  This scale has been associated with good face validity and high levels of convergent validity during exhaustive exercise.16 It consists of an eleven-point (0-10) Likert Scale with verbal anchors of 0, "No Fatigue At All", 1, "Very Small Amount of Fatigue", 2, "Small Amount of Fatigue", 3, "Moderate Fatigue", 4, "Somewhat Fatigued", 5, "Fatigued", 7, "Very Fatigued", 9, "Extremely Fatigued", and 10, "Completely Fatigued"
Perceptual Differences - Changes in Fatigue Scale | Intervention Trial (Day 4) at the 120 minute mark.
  This scale has been associated with good face validity and high levels of convergent validity during exhaustive exercise.16 It consists of an eleven-point (0-10) Likert Scale with verbal anchors of 0, "No Fatigue At All", 1, "Very Small Amount of Fatigue", 2, "Small Amount of Fatigue", 3, "Moderate Fatigue", 4, "Somewhat Fatigued", 5, "Fatigued", 7, "Very Fatigued", 9, "Extremely Fatigued", and 10, "Completely Fatigued"
Perceptual Differences - Changes in Fatigue Scale | Intervention Trial (Day 4) at the 180 minute mark.
  This scale has been associated with good face validity and high levels of convergent validity during exhaustive exercise.16 It consists of an eleven-point (0-10) Likert Scale with verbal anchors of 0, "No Fatigue At All", 1, "Very Small Amount of Fatigue", 2, "Small Amount of Fatigue", 3, "Moderate Fatigue", 4, "Somewhat Fatigued", 5, "Fatigued", 7, "Very Fatigued", 9, "Extremely Fatigued", and 10, "Completely Fatigued"
Perceptual Differences - Changes in Gastrointestinal Distress Scale | Intervention Trial (Day 4) at the -115 minute mark.
  To measure potential gastrointestinal distress or discomfort, a combination of scales will be used including a numeric rating scale (NRS) and the patient's global impression of change (PGIC) scale. The NRS measurement tool has been well psychometrically tested with irritable bowel syndrome (IBS) patients while demonstrating appropriate correlations with GI-symptom severity and excellent construct and discriminant validity for clinical assessments of abdominal pain. This scale will be comprised of a ten-point abdominal pain numeric rating scale with verbal anchors of 1, "None" and 10, "Very Severe".15,23 Furthermore, the PGIC scale has been documented as a commonly used and validated measure of pain. This scale will be comprised of an eight-point Likert scale with verbal anchors of 1, "Very Much Improved", 2, "Much Improved", 3, "Minimally Improved", 4, "No Change", 5, "Minimally Worse", 6, "Much Worse", and 7, "Very Much Worse"
Perceptual Differences - Changes in Gastrointestinal Distress Scale | Intervention Trial (Day 4) at the 0 minute mark.
  To measure potential gastrointestinal distress or discomfort, a combination of scales will be used including a numeric rating scale (NRS) and the patient's global impression of change (PGIC) scale. The NRS measurement tool has been well psychometrically tested with irritable bowel syndrome (IBS) patients while demonstrating appropriate correlations with GI-symptom severity and excellent construct and discriminant validity for clinical assessments of abdominal pain. This scale will be comprised of a ten-point abdominal pain numeric rating scale with verbal anchors of 1, "None" and 10, "Very Severe".15,23 Furthermore, the PGIC scale has been documented as a commonly used and validated measure of pain. This scale will be comprised of an eight-point Likert scale with verbal anchors of 1, "Very Much Improved", 2, "Much Improved", 3, "Minimally Improved", 4, "No Change", 5, "Minimally Worse", 6, "Much Worse", and 7, "Very Much Worse"
Perceptual Differences - Changes in Gastrointestinal Distress Scale | Intervention Trial (Day 4) at the 60 minute mark.
  To measure potential gastrointestinal distress or discomfort, a combination of scales will be used including a numeric rating scale (NRS) and the patient's global impression of change (PGIC) scale. The NRS measurement tool has been well psychometrically tested with irritable bowel syndrome (IBS) patients while demonstrating appropriate correlations with GI-symptom severity and excellent construct and discriminant validity for clinical assessments of abdominal pain. This scale will be comprised of a ten-point abdominal pain numeric rating scale with verbal anchors of 1, "None" and 10, "Very Severe".15,23 Furthermore, the PGIC scale has been documented as a commonly used and validated measure of pain. This scale will be comprised of an eight-point Likert scale with verbal anchors of 1, "Very Much Improved", 2, "Much Improved", 3, "Minimally Improved", 4, "No Change", 5, "Minimally Worse", 6, "Much Worse", and 7, "Very Much Worse"
Perceptual Differences - Changes in Gastrointestinal Distress Scale | Intervention Trial (Day 4) at the 120 minute mark.
  To measure potential gastrointestinal distress or discomfort, a combination of scales will be used including a numeric rating scale (NRS) and the patient's global impression of change (PGIC) scale. The NRS measurement tool has been well psychometrically tested with irritable bowel syndrome (IBS) patients while demonstrating appropriate correlations with GI-symptom severity and excellent construct and discriminant validity for clinical assessments of abdominal pain. This scale will be comprised of a ten-point abdominal pain numeric rating scale with verbal anchors of 1, "None" and 10, "Very Severe".15,23 Furthermore, the PGIC scale has been documented as a commonly used and validated measure of pain. This scale will be comprised of an eight-point Likert scale with verbal anchors of 1, "Very Much Improved", 2, "Much Improved", 3, "Minimally Improved", 4, "No Change", 5, "Minimally Worse", 6, "Much Worse", and 7, "Very Much Worse"
Perceptual Differences - Changes in Gastrointestinal Distress Scale | Intervention Trial (Day 4) at the 180 minute mark.
  To measure potential gastrointestinal distress or discomfort, a combination of scales will be used including a numeric rating scale (NRS) and the patient's global impression of change (PGIC) scale. The NRS measurement tool has been well psychometrically tested with irritable bowel syndrome (IBS) patients while demonstrating appropriate correlations with GI-symptom severity and excellent construct and discriminant validity for clinical assessments of abdominal pain. This scale will be comprised of a ten-point abdominal pain numeric rating scale with verbal anchors of 1, "None" and 10, "Very Severe".15,23 Furthermore, the PGIC scale has been documented as a commonly used and validated measure of pain. This scale will be comprised of an eight-point Likert scale with verbal anchors of 1, "Very Much Improved", 2, "Much Improved", 3, "Minimally Improved", 4, "No Change", 5, "Minimally Worse", 6, "Much Worse", and 7, "Very Much Worse"
Perceptual Differences - Changes in Thermal Sensation Scale | Intervention Trial (Day 4) at the -115 minute mark.
  This scale will be used for the measurement of participant perceptions of heat stress during data collection procedures. The Thermal Sensation Scale is a nine-point (0.0-8.0) Likert Scale with verbal anchors at 0.0, "Unbearably Cold", 1.0, "Very Cold", 2.0, "Cold", 3.0, "Cool", 4.0, "Comfortable", 5.0 "Warm", 6.0, "Hot", 7.0, "Very Hot", and 8.0, "Unbearably Hot"
Perceptual Differences - Changes in Thermal Sensation Scale | Intervention Trial (Day 4) at the 0 minute mark.
  This scale will be used for the measurement of participant perceptions of heat stress during data collection procedures. The Thermal Sensation Scale is a nine-point (0.0-8.0) Likert Scale with verbal anchors at 0.0, "Unbearably Cold", 1.0, "Very Cold", 2.0, "Cold", 3.0, "Cool", 4.0, "Comfortable", 5.0 "Warm", 6.0, "Hot", 7.0, "Very Hot", and 8.0, "Unbearably Hot"
Perceptual Differences - Changes in Thermal Sensation Scale | Intervention Trial (Day 4) at the 60 minute mark.
  This scale will be used for the measurement of participant perceptions of heat stress during data collection procedures. The Thermal Sensation Scale is a nine-point (0.0-8.0) Likert Scale with verbal anchors at 0.0, "Unbearably Cold", 1.0, "Very Cold", 2.0, "Cold", 3.0, "Cool", 4.0, "Comfortable", 5.0 "Warm", 6.0, "Hot", 7.0, "Very Hot", and 8.0, "Unbearably Hot"
Perceptual Differences - Changes in Thermal Sensation Scale | Intervention Trial (Day 4) at the 120 minute mark.
  This scale will be used for the measurement of participant perceptions of heat stress during data collection procedures. The Thermal Sensation Scale is a nine-point (0.0-8.0) Likert Scale with verbal anchors at 0.0, "Unbearably Cold", 1.0, "Very Cold", 2.0, "Cold", 3.0, "Cool", 4.0, "Comfortable", 5.0 "Warm", 6.0, "Hot", 7.0, "Very Hot", and 8.0, "Unbearably Hot"
Perceptual Differences - Changes in Thermal Sensation Scale | Intervention Trial (Day 4) at the 180 minute mark.
  This scale will be used for the measurement of participant perceptions of heat stress during data collection procedures. The Thermal Sensation Scale is a nine-point (0.0-8.0) Likert Scale with verbal anchors at 0.0, "Unbearably Cold", 1.0, "Very Cold", 2.0, "Cold", 3.0, "Cool", 4.0, "Comfortable", 5.0 "Warm", 6.0, "Hot", 7.0, "Very Hot", and 8.0, "Unbearably Hot"
Perceptual Differences - Changes in Thirst Perception Scale | Hydration Baseline Day 1
  A nine-point (1-9) Likert Scale which provides verbal anchors of 1, "Not Thirsty at All"; 3, "A Little Thirsty"; 5, "Moderately Thirsty"; 7, "Very Thirsty"; and 9, "Very, Very Thirsty"
Perceptual Differences - Changes in Thirst Perception Scale | Hydration Baseline Day 2
  A nine-point (1-9) Likert Scale which provides verbal anchors of 1, "Not Thirsty at All"; 3, "A Little Thirsty"; 5, "Moderately Thirsty"; 7, "Very Thirsty"; and 9, "Very, Very Thirsty"
Perceptual Differences - Changes in Thirst Perception Scale | Hydration Baseline Day 3
  A nine-point (1-9) Likert Scale which provides verbal anchors of 1, "Not Thirsty at All"; 3, "A Little Thirsty"; 5, "Moderately Thirsty"; 7, "Very Thirsty"; and 9, "Very, Very Thirsty"
Perceptual Differences - Changes in Thirst Perception Scale | Intervention Trial (Day 4) at the -115 minute mark.
  A nine-point (1-9) Likert Scale which provides verbal anchors of 1, "Not Thirsty at All"; 3, "A Little Thirsty"; 5, "Moderately Thirsty"; 7, "Very Thirsty"; and 9, "Very, Very Thirsty"
Perceptual Differences - Changes in Thirst Perception Scale | Intervention Trial (Day 4) at the 0 minute mark.
  A nine-point (1-9) Likert Scale which provides verbal anchors of 1, "Not Thirsty at All"; 3, "A Little Thirsty"; 5, "Moderately Thirsty"; 7, "Very Thirsty"; and 9, "Very, Very Thirsty"
Perceptual Differences - Changes in Thirst Perception Scale | Intervention Trial (Day 4) at the 60 minute mark.
  A nine-point (1-9) Likert Scale which provides verbal anchors of 1, "Not Thirsty at All"; 3, "A Little Thirsty"; 5, "Moderately Thirsty"; 7, "Very Thirsty"; and 9, "Very, Very Thirsty"
Perceptual Differences - Changes in Thirst Perception Scale | Intervention Trial (Day 4) at the 120 minute mark.
  A nine-point (1-9) Likert Scale which provides verbal anchors of 1, "Not Thirsty at All"; 3, "A Little Thirsty"; 5, "Moderately Thirsty"; 7, "Very Thirsty"; and 9, "Very, Very Thirsty"
Perceptual Differences - Changes in Thirst Perception Scale | Intervention Trial (Day 4) at the 180 minute mark.
  A nine-point (1-9) Likert Scale which provides verbal anchors of 1, "Not Thirsty at All"; 3, "A Little Thirsty"; 5, "Moderately Thirsty"; 7, "Very Thirsty"; and 9, "Very, Very Thirsty"

CONTACTS AND LOCATIONS:
Overall Officials: Douglas J Casa, PhD, Principal Investigator — Korey Stringer Institute - UConn
Locations (1):
- Korey Stringer Institute at the University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No